CLINICAL TRIAL: NCT04561674
Title: The Effect of Web-Based Patient Education on Quality of Life of Patients With Colostomy and Ileostomy: A Randomized Controlled Trial
Brief Title: The Effect of Web-Based Patient Education on Quality of Life of Patients With Colostomy and Ileostomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Collaborators: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Hacer Ozel, Assistant Professor, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 59491012-604.01.02; 31701 (Other: Istanbul University, Cerrahpasa)
Record Dates: First submitted 2020-08-27; First posted 2020-09-23 (Actual); Last update posted 2020-09-23 (Actual); Status verified 2020-09

CONDITIONS: Web Based Patient Education; Quality of Life; Ostomy

STUDY DESIGN:
Intervention Model Description: The study is a randomized controlled experimental research with a pre-test post-test control group design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): The patients in the experimental group participated in "Web-Based Patient Education with Colostomy and Ileostomy" on computer between the third and seventh days after surgery.
  The cards with the website address, username and the website QR code were given to the patients in order to be able to receive education after discharge.The patient and her family received the training from any computer or smartphone connected to the internet.
  Interventions: Other: Implementation of web-based patient education
- Control group (No Intervention): The clinical routine was applied to the control group.

INTERVENTIONS:
Other: Implementation of web-based patient education — Web-Based Patient Education on Colostomy and Ileostomy (WBPECI) was developed in accordance with the principles of the ADDIE instructional design. The web-based education was designed in line with these learning objectives determined. The content of the website was developed in light of the opinions sought from five subject experts. The WBPECI content includes a total of 7 videos, 1 animation with sound, 1 forum and 1 consultation page
  Arms: Experimental Group

SUMMARY:
The purpose of the study is to develop, implement and determine the effects of web-based education programs for patients undergoing colostomy and ileostomy.The study is a randomized controlled experimental research with a pre-test post-test control group design. The study group of the research consisted of individuals, who have an abdominal stoma procedure at a Training and Research Hospital operating under the Ministry of Health in Turkey. 35 individuals were enrolled to the experiment and control groups (N=70). The study group of the hospital was determined as a result of the power analysis performed on an average number of 150 patients, on whom a stoma is opened within a year, with an estimated effect rate of 0.824 and a SD of 0.45, the power being 0.80 and confidence interval p:0.05, as a total of 50 patients, 25 in the experiment group and 25 in the control group. Taking into consideration the data loss that may be experienced, it was planned to enrol 35 individuals to the experiment group and 35 individuals to the control group. The patients were randomly assigned to each group. Homogeneity of patients randomized to the experiment and control groups was checked with a t-test. Research data were collected using an Information Form, Stoma Complications Assessment Form and City of Hope-Quality of Life-Ostomy Questionnaire and Stoma Care Knowledge Assessment Test.

DETAILED DESCRIPTION:
The purpose of the study is to develop, implement and determine the effects of web-based education programs for patients undergoing colostomy and ileostomy.

The study is a randomized controlled experimental research with a pre-test post-test control group design. The study group of the research consisted of individuals, who have an abdominal stoma procedure at a Training and Research Hospital operating under the Ministry of Health in Turkey. 35 individuals were enrolled to the experiment and control groups (N=70). The study group of the hospital was determined as a result of the power analysis performed on an average number of 150 patients, on whom a stoma is opened within a year, with an estimated effect rate of 0.824 and a SD of 0.45, the power being 0.80 and confidence interval p:0.05, as a total of 50 patients, 25 in the experiment group and 25 in the control group. Taking into consideration the data loss that may be experienced, it was planned to enrol 35 individuals to the experiment group and 35 individuals to the control group. The patients were randomly assigned to each group. Homogeneity of patients randomized to the experiment and control groups was checked with a t-test. The stages of the research design were determined completely in accordance with the CONSORT diagram. Data were collected using an Information Form, Stoma Complications Assessment Form and City of Hope-Quality of Life-Ostomy Questionnaire and Stoma Care Knowledge Assessment Test. The study data were analysed with average, standard deviation, frequency, student t test, paired sample t test, variance analysis, Fisher's exact chi-square test, Fisher-Freeman-Halton test and Yates continuity correction test. Significance was assessed at a level of p<0.05.

ELIGIBILITY:
Inclusion Criteria:

Colostomy and ileostomy patients,

* eighteen years and over
* literate
* able to communicate
* who can use computers and internet themselves or their caregivers

Exclusion Criteria:

* under eighteen years
* illiterate
* unable to communicate
* who cannot use computers and the internet themselves or their caregivers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2017-12-18 (Actual); Primary Completion 2018-02-10 (Actual); Study Completion 2018-05-10 (Actual)

PRIMARY OUTCOMES:
Quality of life level | Change from quality of life level at one month
  The City of Hope-Quality of Life-Ostomy Questionnaire was applied to the patients in the experimental."City of Hope-Quality of Life-Ostomy Questionnaire (COH-QOL-OQ)" designed and developed by City of Hope Pain and Palliative Care Resource Centre was first created in 1995 under the name "Quality of life in Cancer Patients".

SECONDARY OUTCOMES:
Stoma Care Knowledge Level | Change from stoma care knowledge level at one day
  Stoma Care Knowledge Assessment Test was applied to the patients in the experimental group.This was prepared in light of the literature in order to assess the patients' level of knowledge on stoma. There are 17 items in the test. An example question is given below: The stool coming out of the stoma causes irritation on the skin surrounding it. The options are true, false and I do not know.

CONTACTS AND LOCATIONS:
Locations (1):
- Saglik Bilimleri Universitesi, Üsküdar, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ang SG, Chen HC, Siah RJ, He HG, Klainin-Yobas P. Stressors relating to patient psychological health following stoma surgery: an integrated literature review. Oncol Nurs Forum. 2013 Nov;40(6):587-94. doi: 10.1188/13.ONF.587-594. PMID 24161637
- [Background] Ambe PC, Kurz NR, Nitschke C, Odeh SF, Moslein G, Zirngibl H. Intestinal Ostomy. Dtsch Arztebl Int. 2018 Mar 16;115(11):182-187. doi: 10.3238/arztebl.2018.0182. PMID 29607805
- [Background] Aquina CT, Iannuzzi JC, Probst CP, Kelly KN, Noyes K, Fleming FJ, Monson JR. Parastomal hernia: a growing problem with new solutions. Dig Surg. 2014;31(4-5):366-76. doi: 10.1159/000369279. Epub 2014 Dec 13. PMID 25531238
- [Background] Barr JE. Assessment and management of stomal complications: a framework for clinical decision making. Ostomy Wound Manage. 2004 Sep;50(9):50-2, 54, 56 passim. PMID 15361633
- [Background] Barrera M Jr, Glasgow RE, McKay HG, Boles SM, Feil EG. Do Internet-based support interventions change perceptions of social support?: An experimental trial of approaches for supporting diabetes self-management. Am J Community Psychol. 2002 Oct;30(5):637-54. doi: 10.1023/A:1016369114780. PMID 12188054
- [Background] Bass SB, Ruzek SB, Gordon TF, Fleisher L, McKeown-Conn N, Moore D. Relationship of Internet health information use with patient behavior and self-efficacy: experiences of newly diagnosed cancer patients who contact the National Cancer Institute's Cancer Information Service. J Health Commun. 2006 Mar;11(2):219-36. doi: 10.1080/10810730500526794. PMID 16537289
- [Background] Berger J, Topp R, Davis L, Jones J, Stewart L. Comparison of Web-based and face-to-face training concerning patient education within a hospital system. J Nurses Staff Dev. 2009 May-Jun;25(3):127-32; quiz 133-4. doi: 10.1097/NND.0b013e3181a56ba0. PMID 19502896
- [Derived] Ozel H, Kaya H. The Effect of Web-Based Patient Education on Quality of Life of Patients With Colostomy and Ileostomy: A Randomized Controlled Trial. J Wound Ostomy Continence Nurs. 2025 Jul-Aug 01;52(4):313-319. doi: 10.1097/WON.0000000000001198. Epub 2025 Jul 24. PMID 40717260